CLINICAL TRIAL: NCT05416840
Title: Effects and Safety of Clonidine Patch on Young and Middle-aged Smokers With Mild Hypertension: a Randomized Controlled Trial (ECLIPSE)
Brief Title: Effects and Safety of Clonidine Patch on Young and Middle-aged Smokers With Mild Hypertension
Acronym: ECLIPSE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jing Liu (Other)
Responsible Party: Sponsor-Investigator, Jing Liu, Director of the Department of Hypertension, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220001
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Hypertension
Keywords: clonidine patch, hypertension, smoking
MeSH Terms: conditions — Hypertension; Smoking | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clonidine (Experimental): Patients will receive clonidine controlled-release patch (2.5 mg), once a week
  Interventions: Drug: Clonidine controlled-release patch
- Amlodipine (Active Comparator): Patients will receive amlodipine (5 mg), once daily
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Clonidine controlled-release patch — Enrolled patients receive clonidine patch (2.5 mg), once a week. The doses are doubled, if the office systolic BP not at goal (<140 mmHg) at 4 weeks.
  All patients receive smoking cessation advice at the beginning, and smoking cessation promotion information is pushed by WeChat three times during the observation period (weeks 2, 4 and 6).
  Arms: Clonidine
Drug: Amlodipine — Enrolled patients receive amlodipine (5 mg), once daily. The doses are doubled, if the office systolic BP not at goal (<140 mmHg) at 4 weeks.
  All patients receive smoking cessation advice at the beginning, and smoking cessation promotion information is pushed by WeChat three times during the observation period (weeks 2, 4 and 6).
  Arms: Amlodipine

SUMMARY:
The optimal antihypertensive treatment strategy in young and middle-aged hypertensive adults remains undefined. Clonidine controlled-release patches administered once a week might have the advantage of convenience. ECLIPSE trial is intended to explore the effect and patient tolerability of clonidine controlled-release patches (one patch per week for a total of 8 weeks) in the treatment of hypertension in young and middle-aged adults, compared with long-acting antihypertensive drug amlodipine. Clonidine patch was demonstrated ameliorating the early withdrawal symptoms during smoking cessation. This trial is also intended to observe its effect on smoking cessation in young and middle-aged male smokers.

DETAILED DESCRIPTION:
The young and middle-aged hypertensive population is growing, but the optimal antihypertensive treatment strategy remains undefined. Young and middle-aged adults have poor adherence to antihypertensive medications and are prone to missed doses, and weekly formulations may be potentially advantageous. As a centrally acting antihypertensive agent, clonidine exerts sustained antihypertensive effects by agonizing alpha2-adrenoceptors. Clonidine controlled-release patches have the advantage of convenience in that they are administered once a week through a transdermal controlled-release technique to achieve a smooth and sustained action of clonidine. However, there is a lack of evidence from clinical trials on its efficacy and tolerability in the treatment of hypertension in young and middle-aged people. ECLIPSE trial is intended to explore the effect and patient tolerability of clonidine controlled-release patches (one patch per week for a total of 8 weeks) in the treatment of hypertension in young and middle-aged adults, compared with long-acting antihypertensive drug amlodipine. Clonidine patch was demonstrated ameliorating the early withdrawal symptoms during smoking cessation and recommended by American Cancer Society to help people quit smoking. Therefore, this trial is also intended to observe its effect on smoking cessation in young and middle-aged male smokers at the same time.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old male with mild hypertension (systolic blood pressure (BP) 140-159 mmHg and/or diastolic BP 90-99 mmHg).
2. History of smoking and a desire to quit.
3. Signed informed consent form.

Exclusion Criteria:

1. History of cardiopulmonary and vascular disease.
2. Severe liver or kidney disease.
3. Night shift workers, drivers, and those who work at height.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — male smokers with mild hypertension
Enrollment: 92 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in clinic sitting systolic BP from baseline at 8-week | 8 weeks
  The change in clinic sitting systolic BP from baseline at 8-week in clonidine group and amlodipine group are analyzed, and between groups difference is compared.

SECONDARY OUTCOMES:
Change in systolic BP in 24 hour ambulatory BP monitoring (ABPM) from baseline at 8-week | 8 weeks
  The change in systolic BP in 24 hour ambulatory BP monitoring (ABPM) from baseline at 8-week in clonidine group and amlodipine group are analyzed, and between groups differences are compared.
Between-group differences in smoking cessation rates at 8-week | 8 weeks
  Between-group differences in smoking cessation rates at 8-week in clonidine group and amlodipine are compared
Drug tolerance and adverse effects during 8 weeks of treatment | 8 weeks
  Drug tolerance and adverse effects during 8 weeks of treatment, clonidine or amlodipine, are analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, MD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No